CLINICAL TRIAL: NCT06440122
Title: The Incidence and Outcomes of Metabolically Active Brown Adipose Tissue (aBAT) in Patients With Pheochromocytoma or Paraganglioma (PPGLs)
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: GafREC-Endo203
Record Dates: First submitted 2024-05-21; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: Brown Adipose Tissue; FDG-PET; Activation; Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with pheochromocytoma or paraganglioma and positive brown adipose tissue on FDG-PET
  Interventions: Diagnostic Test: FDG-PET Scan
- Patients with pheochromocytoma or paraganglioma and negative brown adipose tissue on FDG-PET
  Interventions: Diagnostic Test: FDG-PET Scan

INTERVENTIONS:
Diagnostic Test: FDG-PET Scan — Positive for activated brown adipose tissue (SUVmax >1.5) FDG-PET scan

SUMMARY:
White adipose tissue (WAT) and brown adipose tissue (BAT) form the main adipose tissue subtypes in humans and several animals. BAT, owing to its unique metabolic function, has been of increased focus and interest in metabolic research (1). BAT forms the major organ of non-shivering thermogenesis in the body, and is dependent on the large concentration of mitochondria and increased uncoupling protein-1 (UCP-1) activity present in this type of tissue (2). There are numerous triggers for the metabolic activation of BAT including cold temperature, low body mass index (BMI), adrenergic agonists, and elevated concentration of thyroid hormones (3).

BAT is found more abundantly in fetuses and infants, with significant regression into adulthood. The main areas where BAT can be found are the neck, mediastinum, axilla, retroperitoneum, and abdominal wall (4). Clinical research suggests that activation and thermogenesis in BAT are mediated by noradrenaline release from the sympathetic nervous system (5). With the increasing use of fluorodeoxyglucose positron emission tomography (18FDG-PET) imaging, there has been an increased detection rate of activated brown adipose tissue (aBAT); this may affect diagnoses and lead to false-positive reporting (6).

Phaeochromocytomas/paragangliomas (PPGLs) are chromaffin-cell-derived endocrine tumors that emerge from the adrenal medulla or extra-adrenal ganglia. High FDG accumulation has been commonly noted in aBAT in patients with catecholamine-producing tumours, with subsequent resolution of these findings after resection of the tumour (7). This finding is likely related to the increased glucose transport related to noradrenaline excess (4). BAT has traditionally been considered to mainly express β3-adrenoreceptors; however, in vitro studies have indicated that activated β2-adrenoreceptors may be the main driving force behind thermogenesis (8).

Studies reviewing PPGLs have shown an aBAT detection rate of 7.8% to 42.8% on FDG-PET imaging, correlating with elevated catecholamine levels but without clear correlation to germline mutations (9-12). In one study, this imaging finding was associated with a statistically significant reduction in overall survival (12). Standardisation for the 'standardised uptake value' (SUV) cut-offs for aBAT on FDG-PET are lacking, but these are often reported between 1.0 and 2.0 (13); in previous studies of PPGL, a cut-off value of >1.5 has been employed (10, 12).

Research on the clinical implications of aBAT in patients with PPGL remains scarce. The main objectives of this study were to gain further insights into BAT activation rates in patients with PPGLs and how this may relate to patient demographics, biochemistry, radiological features, mutational status, and outcomes. The main hypotheses were that aBAT rates would be significantly linked to the severity of catecholamine excess and could be considered a poor prognostic feature.

DETAILED DESCRIPTION:
References:

1. Santhanam P, Solnes L, Hannukainen JC, Taïeb D. Adiposity-related cancer and functional imaging of brown adipose tissue. Endocr Pract. 2015;21(11):1282-90.
2. Fenzl A, Kiefer FW. Brown adipose tissue and thermogenesis. Horm Mol Biol Clin Investig. 2014;19(1):25-37.
3. Marlatt KL, Ravussin E. Brown adipose tissue: An update on recent findings. Curr Obes Rep. 2017;6(4):389-96.
4. Iyer RB, Guo CC, Perrier N. Adrenal pheochromocytoma with surrounding brown fat stimulation. AJR Am J Roentgenol. 2009;192(1):300-1.
5. Bartness TJ, Vaughan CH, Song CK. Sympathetic and sensory innervation of brown adipose tissue. Int J Obes (Lond). 2010;34 Suppl 1(S1):S36-42.
6. Nedergaard J, Bengtsson T, Cannon B. Unexpected evidence for active brown adipose tissue in adult humans. Am J Physiol Endocrinol Metab. 2007;293(2):E444-52.
7. Terada E, Ashida K, Ohe K, Sakamoto S, Hasuzawa N, Nomura M. Brown adipose activation and reversible beige coloration in adipose tissue with multiple accumulations of 18F-fluorodeoxyglucose in sporadic paraganglioma: A case report. Clin Case Rep. 2019;7(7):1399-403.
8. Blondin DP, Nielsen S, Kuipers EN, Severinsen MC, Jensen VH, Miard S, et al. Human brown adipocyte thermogenesis is driven by β2-AR stimulation. Cell Metab. 2020;32(2):287-300.e7.
9. Wang Q, Zhang M, Ning G, Gu W, Su T, Xu M, et al. Brown adipose tissue in humans is activated by elevated plasma catecholamines levels and is inversely related to central obesity. PLoS One. 2011;6(6):e21006.
10. Puar T, van Berkel A, Gotthardt M, Havekes B, Hermus ARMM, Lenders JWM, et al. Genotype-dependent brown adipose tissue activation in patients with pheochromocytoma and paraganglioma. J Clin Endocrinol Metab. 2016;101(1):224-32.
11. Hadi M, Chen CC, Whatley M, Pacak K, Carrasquillo JA. Brown fat imaging with (18)F-6-fluorodopamine PET/CT, (18)F-FDG PET/CT, and (123)I-MIBG SPECT: a study of patients being evaluated for pheochromocytoma. J Nucl Med. 2007;48(7):1077-83.
12. Abdul Sater Z, Jha A, Hamimi A, Mandl A, Hartley IR, Gubbi S, et al. Pheochromocytoma and paraganglioma patients with poor survival often show brown adipose tissue activation. J Clin Endocrinol Metab. 2020;105(4):1176-85.
13. Sampath SC, Sampath SC, Bredella MA, Cypess AM, Torriani M. Imaging of brown adipose tissue: State of the art. Radiology. 2016;280(1):4-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed pheochromocytoma or paraganglioma who have undergone a FDG-PET as part of staging process.

Exclusion Criteria:

* Patients with any other neoplasm other than pheochromocytoma or paraganglioma

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patients with confirmed pheochromocytoma or paraganglioma treated at King's College Hospital NHS Foundation Trust Endocrinology department who underwent an FDG-PET scan.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with pheochromocytoma and metabolically active brown adipose tissue on FGD-PET scan | through study completion, an average of 1 year
Number of patients with paraganglioma and metabolically active brown adipose tissue on FGD-PET scan | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Metabolically active brown adipose tissue and presence of germ-line mutations (NHL) in patients with pheochromocytoma and paraganglioma | through study completion, an average of 1 year
  We are going to assess if patients with metabolically active adipose tissue and pheochromocytoma or paraganglioma present with germ-line mutations (VHL) or whether this occurs in patients with sporadic tumours
Metabolically active brown adipose tissue and presence of germ-line mutations (NF-1) in patients with pheochromocytoma and paraganglioma | through study completion, an average of 1 year
  We are going to assess if patients with metabolically active adipose tissue and pheochromocytoma or paraganglioma present with germ-line mutations (NF-1) or whether this occurs in patients with sporadic tumours
Metabolically active brown adipose tissue and presence of germ-line mutations (MEN) in patients with pheochromocytoma and paraganglioma | through study completion, an average of 1 year
  We are going to assess if patients with metabolically active adipose tissue and pheochromocytoma or paraganglioma present with germ-line mutations (MEN) or whether this occurs in patients with sporadic tumours

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Dimitriadis, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom of Great Britain and Northern Ireland, United Kingdom

REFERENCES:
- [Background] Santhanam P, Solnes L, Hannukainen JC, Taieb D. ADIPOSITY-RELATED CANCER AND FUNCTIONAL IMAGING OF BROWN ADIPOSE TISSUE. Endocr Pract. 2015 Nov;21(11):1282-90. doi: 10.4158/EP15870.RA. Epub 2015 Aug 17. PMID 26280202
- [Background] Fenzl A, Kiefer FW. Brown adipose tissue and thermogenesis. Horm Mol Biol Clin Investig. 2014 Jul;19(1):25-37. doi: 10.1515/hmbci-2014-0022. PMID 25390014
- [Background] Marlatt KL, Ravussin E. Brown Adipose Tissue: an Update on Recent Findings. Curr Obes Rep. 2017 Dec;6(4):389-396. doi: 10.1007/s13679-017-0283-6. PMID 29101739
- [Background] Iyer RB, Guo CC, Perrier N. Adrenal pheochromocytoma with surrounding brown fat stimulation. AJR Am J Roentgenol. 2009 Jan;192(1):300-1. doi: 10.2214/AJR.08.1166. No abstract available. PMID 19098214
- [Background] Bartness TJ, Vaughan CH, Song CK. Sympathetic and sensory innervation of brown adipose tissue. Int J Obes (Lond). 2010 Oct;34 Suppl 1(0 1):S36-42. doi: 10.1038/ijo.2010.182. PMID 20935665
- [Background] Nedergaard J, Bengtsson T, Cannon B. Unexpected evidence for active brown adipose tissue in adult humans. Am J Physiol Endocrinol Metab. 2007 Aug;293(2):E444-52. doi: 10.1152/ajpendo.00691.2006. Epub 2007 May 1. PMID 17473055
- [Background] Terada E, Ashida K, Ohe K, Sakamoto S, Hasuzawa N, Nomura M. Brown adipose activation and reversible beige coloration in adipose tissue with multiple accumulations of 18F-fluorodeoxyglucose in sporadic paraganglioma: A case report. Clin Case Rep. 2019 Jun 11;7(7):1399-1403. doi: 10.1002/ccr3.2259. eCollection 2019 Jul. PMID 31360497
- [Background] Blondin DP, Nielsen S, Kuipers EN, Severinsen MC, Jensen VH, Miard S, Jespersen NZ, Kooijman S, Boon MR, Fortin M, Phoenix S, Frisch F, Guerin B, Turcotte EE, Haman F, Richard D, Picard F, Rensen PCN, Scheele C, Carpentier AC. Human Brown Adipocyte Thermogenesis Is Driven by beta2-AR Stimulation. Cell Metab. 2020 Aug 4;32(2):287-300.e7. doi: 10.1016/j.cmet.2020.07.005. PMID 32755608
- [Background] Wang Q, Zhang M, Ning G, Gu W, Su T, Xu M, Li B, Wang W. Brown adipose tissue in humans is activated by elevated plasma catecholamines levels and is inversely related to central obesity. PLoS One. 2011;6(6):e21006. doi: 10.1371/journal.pone.0021006. Epub 2011 Jun 20. PMID 21701596
- [Background] Puar T, van Berkel A, Gotthardt M, Havekes B, Hermus AR, Lenders JW, van Marken Lichtenbelt WD, Xu Y, Brans B, Timmers HJ. Genotype-Dependent Brown Adipose Tissue Activation in Patients With Pheochromocytoma and Paraganglioma. J Clin Endocrinol Metab. 2016 Jan;101(1):224-32. doi: 10.1210/jc.2015-3205. Epub 2015 Nov 17. PMID 26574955
- [Background] Hadi M, Chen CC, Whatley M, Pacak K, Carrasquillo JA. Brown fat imaging with (18)F-6-fluorodopamine PET/CT, (18)F-FDG PET/CT, and (123)I-MIBG SPECT: a study of patients being evaluated for pheochromocytoma. J Nucl Med. 2007 Jul;48(7):1077-83. doi: 10.2967/jnumed.106.035915. Epub 2007 Jun 15. PMID 17574980
- [Background] Abdul Sater Z, Jha A, Hamimi A, Mandl A, Hartley IR, Gubbi S, Patel M, Gonzales M, Taieb D, Civelek AC, Gharib AM, Auh S, O'Mara AE, Pacak K, Cypess AM. Pheochromocytoma and Paraganglioma Patients With Poor Survival Often Show Brown Adipose Tissue Activation. J Clin Endocrinol Metab. 2020 Apr 1;105(4):1176-85. doi: 10.1210/clinem/dgz314. PMID 31903484
- [Background] Sampath SC, Sampath SC, Bredella MA, Cypess AM, Torriani M. Imaging of Brown Adipose Tissue: State of the Art. Radiology. 2016 Jul;280(1):4-19. doi: 10.1148/radiol.2016150390. PMID 27322970